CLINICAL TRIAL: NCT05424094
Title: Health-related Quality of Life in Overweight and Obese Children/Adolescents - a Pilot Project in the 'Kinderleicht' Group Programme
Brief Title: HRQoL in Overweight and Obese Children/Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Frank Wieber (Other)
Responsible Party: Sponsor-Investigator, Frank Wieber, professor doctor Frank Wieber, Zurich University of Applied Sciences
Organization: Zurich University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRQoL_29.12.21
Record Dates: First submitted 2021-11-25; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Obesity, Childhood; Health Related Quality of Life; Intervention Program; Obesity, Adolescent; Overweight and Obesity
Keywords: obesity; overweight; health related quality of life
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 'kinderleicht' programme (Experimental): Children receive coaching in the areas of behaviour, exercise, nutrition and medicine from qualified professionals.
  Interventions: Behavioral: multi-professional group programme 'kinderleicht'

INTERVENTIONS:
Behavioral: multi-professional group programme 'kinderleicht' — 12-16 children/adolescents who participate in the multi-professional group programme 'kinderleicht' receive coaching in the areas of behaviour, exercise, nutrition and medicine from qualified professionals on fridays during 11 months.

SUMMARY:
The primary aim of the present study is to record changes in the health-related quality of life (HRQoL) of children/adolescents participating in the multi-professional group programme 'kinderleicht' in 2022 over the course of the eleven-month active phase. In addition, these data will be examined for correlation with changes in BMI, waist and hip circumference, and motor performance.

Secondarily, the study addresses the questions of whether the recording of HROoL by means of the KINDL questionnaire is practicable for the programme leaders and what benefit can be gained from the analysed data for future cohorts.

DETAILED DESCRIPTION:
According to the 2021 publication of the WHO European Childhood Obesity Surveillance Initiative (COSI), overweight and obesity in children and adolescents remains one of the most serious health problems facing the European population in the 21st century. The WHO responded to this problem in 2019 with a review paper on the propagated intervention approaches. With its developed national guidelines, Switzerland relies on multiprofessional group programmes. One of the eleven currently tested and certified programmes is 'kinderleicht' in Chur. The nationwide KIDSSTEP study from 2014 - on which the nationwide guidelines for multiprofessional group programmes are based - shows that it is imperative to record the health-related quality of life (HRQoL) of the children and adolescents as well as their families. In practice, however, this evidence is still too little implemented. Using the example of 'kinderleicht', it is to show that the recording and documentation of HRQoL is practicable and can provide valuable insights for both programme participants and programme managers. The primary goal is to record the health-related quality of life of children and adolescents participating in the multi-professional group programme 'kinderleicht' in 2022 over the course of the eleven-month active phase. At the same time, these data are to be correlated and interpreted with changes in BMI, waist and hip circumference and motor performance. Secondarily, possible sensitive/difficult phases of a participant during the active phase of the intervention will be identified in order to provide the best possible coaching to the families of future cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. girls/boys aged 7-17 years.
2. participation with children
3. age-adjusted BMI: P > 97th percentile or 90th-97th percentile + diseases whose prognosis is worsened by the overweight or are the result of the overweight
4. medical examination unobjectionable
5. motivation to participate in the programme is given
6. written informed consent of the participant, 6.1. for children up to 14 years of age, verbal consent of the child is sufficient, plus written consent of the parents or a legal representative 6.2. for adolescents aged 14 and over, written consent from the adolescent is sufficient.

Exclusion Criteria:

1. BMI < 90 percentile
2. not part of 'easy for children
3. medical examination questionable
4. no motivation to participate in the programme
5. no verbal and/or written consent of the children and their parents/legal representatives

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
health related quality of life (HRQoL) over 11 months | 11 months
  measured with the 'KINDL'-questionair; linkert scaled with a maximum value of 100 and a minimum value of 0 (points); the higher the score the better

SECONDARY OUTCOMES:
Rate of Body Mass Index (BMI) over 11 months | 11 months
  weight (kilograms) and height (meters) will be combined to report the BMI rate in kg/m^2; the BMI rate is age-appropriate for children and adolescents; the aim of the intervention programme is to reduce the BMI rate in obese children so a lower BMI rate is better than a higher one
hip-waist ratio | 11 months
  hip and waist circumference in centimetres are combined to hip-waist ratio
motor performance | 11 months
  motor performance ist measured in seven categories by test DKT-Fitnessolympiade; Results are graded according to the German school grading system; minimum grade 6 and maximum grade 1; the lower the grade the better

IPD SHARING:
Plan to Share IPD: No